CLINICAL TRIAL: NCT05666076
Title: Ultrasound-guided Shoulder PENG Block Versus Suprascapular Nerve Block for Postoperative Analgesia in Shoulder Arthroscopy; A Prospective Randomized Controlled Study
Brief Title: Peng Block or Suprascapular Nerve Block for Postoperative Analgesia in Shoulder Artroscopy ?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gokhan Sertcakacilar, MD, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022-360
Record Dates: First submitted 2022-11-28; First posted 2022-12-27 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Orthopedic Disorder; Shoulder Pain; Surgery; Analgesia
Keywords: peng block; suprascapular nerve block; postoperative analgesia
MeSH Terms: conditions — Musculoskeletal Diseases; Shoulder Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PENG (Active Comparator): The investigators performed a pericapsular nerve block on that patient group for postoperative analgesia.
  Interventions: Procedure: Pericapsular nerve block; Drug: Bupivacaine Hydrochloride
- Group SSNB (Active Comparator): The investigators performed a suprascapular nerve block on that patient group for postoperative analgesia.
  Interventions: Procedure: Suprascapular nerve block; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Procedure: Pericapsular nerve block — The investigators will perform a pericapsular nerve block on that patient group for postoperative analgesia in shoulder arthroscopy.
  Arms: Group PENG
Procedure: Suprascapular nerve block — The investigators will perform a suprascapular nerve block on that patient group for postoperative analgesia in shoulder arthroscopy.
  Arms: Group SSNB
Drug: Bupivacaine Hydrochloride — The investigators will perform a pericapsular nerve block on that patient group for postoperative analgesia with bupivacaine hydrochloride
  Arms: Group PENG
Drug: Bupivacaine Hydrochloride — The investigators will perform a suprascapular nerve block on that patient group for postoperative analgesia with bupivacaine hydrochloride
  Arms: Group SSNB

SUMMARY:
Arthroscopic shoulder surgery, which has been frequently applied in recent years, provides long-term positive clinical results and increases the quality of life after surgery, while it can cause severe pain in the early postoperative period. Postoperative pain management is very important in shoulder arthroplasty. Adequate pain control; mental state, nutrition, cost of care, rehabilitation, and patient satisfaction, are of great importance for the patients' recovery and contribute to a successful surgical outcome.

In this study, the investigators aimed to compare the effects of suprascapular nerve block and shoulder pericapsular nerve block, which will be performed preoperatively with ultrasound, on the level of postoperative pain in patients who will undergo shoulder arthroscopy surgery under general anesthesia.

DETAILED DESCRIPTION:
As a result of the power analysis the investigators conducted for this study, the minimum sample size was calculated as 32 people for each group, 64 people in total, at the 90% confidence interval.

64 patients who meet the inclusion criteria will be included in our study. The participants will be randomized and divided into 2 groups. Accordingly, the PENG block will be applied to 32 patients, and the suprascapular block will be applied to 32 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will have shoulder arthroscopy surgery under general anesthesia
* Ages of 18-75
* ASA I-III

Exclusion Criteria:

* Patients with deformity and pathology in the shoulder region
* Patients with known local anesthetic allergy
* Patients with BMI>35
* Patients with alcohol and substance addiction
* Patients with opioid addiction
* Patients who cannot perceive and evaluate pain, such as psychiatric illness, mental retardation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of the study is the patients' postoperative pain scores (NRS) | 36 hours postoperatively
  Numerical rating scale (NRS) at 1, 6, 12, 18, 24, 30, and 36th hours. A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
Postoperative 36-hour total tramadol hydrochloride consumption | 36 hours postoperatively
  This will be measured by the PCA device in the 36 hours after

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
From the date of publication, available data may begin. If requested, the data will be shared with the anesthetists dealing with shoulder blocks.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Two year within the publication date.

REFERENCES:
- [Background] Sun C, Zhang X, Ji X, Yu P, Cai X, Yang H. Suprascapular nerve block and axillary nerve block versus interscalene nerve block for arthroscopic shoulder surgery: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2021 Nov 5;100(44):e27661. doi: 10.1097/MD.0000000000027661. PMID 34871240
- [Background] Kupeli I, Yazici Kara M. Anesthesia or analgesia? New block for shoulder surgery: pericapsular nerve group block. Braz J Anesthesiol. 2022 Sep-Oct;72(5):669-672. doi: 10.1016/j.bjane.2021.05.009. Epub 2021 Jun 9. PMID 34118263